CLINICAL TRIAL: NCT02211807
Title: The Risk of Suicidality and Suicide Attempt Among HIV Patients Initiating Efavirenz-containing Versus Efavirenz-free Antiretroviral Regimens
Brief Title: Suicidality and Suicide Attempt Among HIV Patients on Efavirenz-containing Versus Efavirenz-free Antiretroviral Regimens
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Truven Health Analytics (Unknown)
Responsible Party: Sponsor
Other Study IDs: AI266-960
Record Dates: First submitted 2014-07-21; First posted 2014-08-08 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients initiating an Efavirenz: Patients initiating an Efavirenz-containing antiretroviral regimen
- Patients initiating an Efavirenz-free regimen

SUMMARY:
The purpose of this study was to compare the frequency of suicidality and suicide attempt among HIV patients starting treatment with Efavirenz and with patients starting treatment with other HIV medications.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* At least 6 months of enrollment before first prescription
* Antiretroviral naive

Exclusion Criteria:

* No diagnosis of HIV on patient record
* Age < 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in a commercial insurance database and a Medicaid database
Sampling Method: Probability Sample
Enrollment: 11400 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of cases of Suicidality, defined as suicidal ideation and suicide attempt | Patients will be followed from date of index fill of efavirenz or comparator antiretrovirals until earliest of date of suicidality claim,30th day after the last day of the days supply of the index medication,last day of enrollment or end of study period

SECONDARY OUTCOMES:
Number of suicide attempt cases, defined as an inpatient or emergency room claim with at least one ICD-9-CM code for suicide attempt | Patients will be followed from date of index fill of efavirenz or comparator antiretrovirals until earliest of date of suicidality claim,30th day after the last day of the days supply of the index medication,last day of enrollment or end of study period
Number of suicide attempt cases | Patients will be followed from date of index fill of efavirenz or comparator antiretrovirals until earliest of date of suicidality claim,30th day after the last day of the days supply of the index medication,last day of enrollment or end of study period
  Expanded definition, defined as an inpatient of emergency department claim for suicidal attempt or a claim for toxic effects of poisoning, open wound to elbow, wrist or forearm, of asphyxiation plus a diagnosis of psychiatric disorders

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx